CLINICAL TRIAL: NCT06581068
Title: Automation of the In Vitro Fertilization Laboratory: A Validation Study
Brief Title: Automation of the In Vitro Fertilization Laboratory
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Conceivable Life Sciences (Industry)
Collaborators: Hope Fertility Center (Unknown); Reina Madre (Unknown); Nascere (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRC-IN-017
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Infertility; ART
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AURA assisted ART treatment (Experimental): The laboratory element of the patient's ART treatment will be automated through the use of the AURA device. This includes sperm preparation and egg retrieval from follicular fluid. 1 out of every 4 eggs will be randomly removed from the AURA system and treated by standard care. The remaining eggs will be maintained in the AURA system and further processed automatically for egg denudation, fertilization, embryo culture, embryo cryopreservation.
  Interventions: Device: AURA assisted ART treatment

INTERVENTIONS:
Device: AURA assisted ART treatment — The AURA device consists of five subsystems, which will operate in logical sequence to deliver comprehensive automation of the laboratory element of an ART cycle. The AURA treatment begins after ovarian stimulation, on the day of egg collection. A sperm sample is provided on the same day of egg collection. Sperm samples will be prepared by the C:SPERM subsystem. Follicular fluid obtained at egg collection will be processed by the C:EGG subsystem. 3 out of every 4 cumulus-oocyte complexes (COCs) recovered will be denuded by the C:EGG subsystem. These denuded eggs will be fertilized by the C:ICSI subsystem, incubated in the C:CULTURE subsystem and all resulting suitable embryos will be vitrified by the C:VIT subsystem. Thawed embryos may be used in conventional frozen embryo transfers.

SUMMARY:
Enrolled patients will undergo an Assisted Reproductive technology (ART) treatment using intracytoplasmic sperm injection (ICSI, the direct injection of a single sperm cell into an oocyte) as the method of insemination. In this prospective cohort study, patients' sperm, eggs, and embryos will be processed using an automated system called AURA (Conceivable Life Sciences), which consists of five subsystems. Specifically, sperm samples will be prepared for fertilization using the subsystem C:SPERM. Cumulus-oocyte complexes (COCs) containing the oocytes will be isolated from follicular fluid using the subsystem C:EGG. One out of every four COCs will be removed from the AURA system at random and processed according to the local treatment clinic's standard operating procedure. All other COCs will continue automated procedures and will be denuded, fertilized, incubated, and vitrified using the AURA subsystems C:EGG. C:ICSI, C:CULTURE and C:VIT, respectively. All automated procedures will be conducted under the supervision of a laboratory manager, who can intervene, address any potential anomalies, and override any steps undertaken by the automated AURA system. The study aims to deliver a descriptive evaluation of the AURA system, including assessing the device's performance, defined by its level of automation, efficiency, and throughput. As a secondary objective, the study aims to characterize the clinical performance of each of AURA's subsystems and correlate this performance against pre-established benchmarks in a non-inferiority statistical analysis. Finally, the study seeks to collect technical data related to AURA's hardware and software operation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the patients before treatment.
* Medical indication to perform assisted reproductive technology.
* Body mass index between 20 and 29 kg/m2 (female participants only).
* For women with indication of utilizing autologous eggs:

  * Anti-Müllerian Hormone (AMH) value of at least 1.5 ng/mL.
  * 18 - 39 years of age.
* For women utilizing donor eggs (egg donor age 18-28 years):

  * 18 - 45 years of age.

Exclusion Criteria:

* Patients diagnosed with recurrent pregnancy loss.
* Inaccessible ovaries for puncture.
* History of total or partial fertilization failure in a previous fertility treatment.
* History of repeated implantation failure defined as three previous unsuccessful embryo transfers.
* Uterine factors (e.g. fibroids, uterine surgeries, Müllerian malformations) at the discretion of the medical team and based on its impact on success and/or risk to the patient or the pregnancy may compromise treatment prognosis).
* Untreated hydrosalpinx
* Severe endometriosis III, IV, presence of endometriomas and/or history of endometrioma resection.
* Polycystic ovarian syndrome.
* Patients with any of the following severe male factor infertility:

  * Sperm concentrations less than 5 million per mL
  * Progressive motility less than 5%
  * Others (e.g, globozoospermia and seminal infections) at the discretion of the medical team and based on its impact on success.
  * Surgically retrieved sperm (TESE, MESA, PESA)
* Pre-existing conditions compromising reproductive (e.g., thrombophilia, chronic degenerative and autoimmune diseases, uncontrolled hormonal disorders).
* Any other case of abnormalities that could compromise success rates according to the criteria of clinical personnel in charge.
* Inability to adhere to the medical protocols and/or schedules for personal reasons.
* Intercurrent medical disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Autonomy | 9 months
  proportion of tasks successfully completed by the AURA system without requiring human intervention.
Procedural timings | 9 months
  time employed by the AURA system to complete each of its automated tasks.

SECONDARY OUTCOMES:
Sperm motility post preparation | 9 months
  proportion of sperm cells displaying motility (progressive) following sperm preparation.
Denudation survival rate | 9 months
  proportion of oocytes that do not lyse or degenerate at the end of automated egg discovery and denudation.
ICSI damage rate | 9 months
  Proportion of oocytes that lyse or degenerate within 24 hours after ICSI.
Normal fertilization rate | 9 months
  proportion of oocytes with two pronuclei (and two polar bodies if assessable) 16 hrs after ICSI.
Blastocyst development rate | 9 months
  proportion of embryos with expanded/expanding blastocoele and discernible inner cell mass (ICM) and trophectoderm (TE) observed on day 5 of development (where ICSI is performed on Day 0) as a function of normally fertilized oocytes.
Usable blastocyst development rate | 9 months
  proportion of blastocysts of sufficient quality for transfer or cryopreservation observed within 6 days of fertilization as a function of mature (MII) eggs injected with sperm during ICSI.
Blastocyst cryosurvival rate | 9 months
  proportion of cryopreserved blastocysts that present re-expansion within 2 hours of warming.
Implantation rate | 9 months
  number of gestational sacs detected by ultrasound scan performed at gestation weeks 5-8 per total number of embryos transferred.
Clinical pregnancy rate | 9 months
  number of patients with fetal heartbeats detected by ultrasound scan performed at gestation weeks 5-8 per total number of patients with an embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Cohen, PhD, Principal Investigator — Conceivable Life Sciences
Locations (2):
- Mexico (2):
  - New Hope Fertility Centre, Mexico City, Mexico City, Mexico City
  - Reina Madre, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. Proposals should be directed to Jacques@Conceivable.life; to gain access, data requestors will need to sign a data access agreement.